CLINICAL TRIAL: NCT01797952
Title: A Randomized Double Blind Placebo Controlled Phase III Study of Efficacy of Lactobacillus CD2 Lozenges in Preventing High-Dose Chemotherapy Induced Oral Mucositis in Patients Undergoing Myeloablative Hematopoietic Stem Cell Transplantation
Brief Title: A Phase III Study of Efficacy of Lactobacillus CD2 Lozenges in Preventing High-Dose Chemotherapy Induced Oral Mucositis in Patients Undergoing Myeloablative Hematopoietic Stem Cell Transplantation
Acronym: mucositis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI was away on sabbatical for 2 years.Protocol is being revised before starting the study.
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Atul Sharma, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P 1201
Record Dates: First submitted 2013-02-19; First posted 2013-02-25 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Oral Mucositis in Patients Undergoing HSCT
Keywords: lactobacillus CD 2; oral mucositis; hematopoietic stem cell transplantation
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus CD 2 lozenges (Active Comparator): 2x109 (2 billion) viable cells of Lactobacillus CD2 as active ingredient
  Interventions: Drug: Lactobacillus CD 2; Other: Placebo
- Placebo lozenges (Placebo Comparator): The placebo is a mix of sugars and salts used as excipients in the active formulation
  Interventions: Drug: Lactobacillus CD 2; Other: Placebo

INTERVENTIONS:
Drug: Lactobacillus CD 2 — 2x109 (2 billion) viable cells of Lactobacillus CD2 as active ingredient
Other: Placebo — The placebo is a mix of sugars and salts used as excipients in the active formulation

SUMMARY:
The study will be conducted at departments of Medical Oncology and Hematology, All India Institute of Medical Sciences (AIIMS).

Patients with various malignancies who are taken up for high dose chemotherapy followed by stem cells transplant (blood and marrow transplant) have very high chances of developing severe oral mucositis (generally 60-80% in different studies and our own previous experiences). This not only causes significant morbidity but also hampers quality of life needing use of parenteral nutrition, analgesics, and antibiotics.

No definite treatment exists for prevention or treatment of oral mucositis in this group of patients. Though one study has suggested that use of IV palifermin (a keratinocyte growth factor) will reduce duration and severity. Palifermin is very expensive and not available in country. Recently investigators have shown effectiveness of a probiotic Lactobacillus CD 2 in reducing incidence and severity of chemo-radiotherapy induced mucositis in head and neck squamous cell cancer patients. (Published online in European Journal of Cancer: http://dx.doi.org/10.1016/j.ejca.2011.06.010)European Journal of Cancer 2012;4:875-881.No significant toxicity has been reported with its use.

A pilot study on similar aspect was completed recently at our center(Clinical trial.gov identifier:NCT 01480011) and in 31 patients who received this only 6 (20%) developed grade III or IV Mucositis. Now, investigators want to study the efficacy of this drug to reduce severity of mucositis in patients undergoing myeloablative hematopoietic stem cell transplantation. The study drug and placebo will be supplied by CD Pharma India Private Limited.

Investigators further give undertaking that study will be carried as per GCP and declaration of Helsinki.

DETAILED DESCRIPTION:
Study Design Placebo controlled double blind randomized, multi center clinical trial.

Study Population and Number of Subjects Total of 108 patients undergoing myeloablative allogeneic or autologous hematopoietic stem cell transplantation and receiving high-dose chemotherapy as conditioning regimen at AIIMS (departments of Medical Oncology and Hematology) will be enrolled for the study and will be equally divided in two groups (drug and placebo).

Study Center The study will be carried at Departments of Medical Oncology and Hematology of All India Institute of Medical Sciences, New Delhi, India.

More centers are likely to be added.

Study Objectives To test whether the probiotic Lactobacillus CD2 (drug) lozenges can reduce the incidence and severity of conditioning therapy induced oral mucositis in patients undergoing haematopoietic stem cell transplantation.

Investigational Product Drug: The trial medication is in the form of lozenge, which is supposed to be dissolved by itself in mouth.

It contains not less than 2x109 (2 billion) viable cells of Lactobacillus CD2 as active ingredient.

Placebo: The placebo is a mix of sugars and salts used as excipients in the active formulation.

Note: Placebo and drug lozenges will be similar in physical appearance and color.

Dose of Study drug The daily dose of trial medications will be 4-6 lozenges per day, one lozenge to be taken every 2-3 hours preferably not before the meal. The lozenge should be kept in mouth for it to dissolve by itself. A hot beverage (e.g. tea, coffee, milk etc.) should not be taken for at least half an hour before and after the medication since elevated temperature can inactivate the bacteria.

Duration of treatment The treatment will start 4-7 days before starting chemotherapy for conditioning regime of HSCT and will continue till resolution of mucositis or Day+24 post stem cell infusion which-ever is earlier.

Efficacy Assessments

Clinical activity will be defined as reduction in the incidence and severity of chemotherapy induced mucositis in HSCT patients. Most recent version of CTCAE; clinical score of CTC V4.03 ( as also outlined in CTCAE version 3.0) will be used for mucositis assessment. Also,WHO and Oral Mucositis assessment score will be recorded. The study will have the following primary and secondary endpoints:

Primary endpoint

1. Determine the incidence of grade III and IV mucositis in patients undergoing allogeneic or autologous haematopoietic stem cell transplantation in two groups.

Secondary endpoint

1. Determine the incidence of all Grade of mucositis in patients undergoing allogenic or autologous haematopoietic stem cell transplantation in two groups.
2. Duration of and time period for healing of chemotherapy induced oral mucositis.
3. Determine incidence and severity of dysphagia and requirement of IV antibiotics in two groups

Safety Assessments

1. Medical History
2. Physical Examination
3. Vital Signs (blood pressure, pulse rate and respiratory rate)
4. Laboratory Examinations
5. Adverse Events

ELIGIBILITY:
Inclusion Criteria:

1. Age between 10 and 70 years.
2. Karnofsky Performance Score ≥ 70%.
3. Confirmed histological diagnosis of cancer/leukaemia for which haematopoietic stem cell transplantation is as approved modality of therapy.
4. Patients eligible to receive high-dose chemotherapy as part of conditioning regime.
5. Concomitant co morbid condition if present, controlled by medicines.
6. Serum creatinine upto 1.8mg/dl.
7. Total bilirubin 2mg/dl.
8. Liver enzymes within three times of normal limit.
9. Expected survival > 6 months.

Exclusion Criteria:

1. Pregnant women and lactating mothers.
2. Patients with history of AIDS
3. Patients who have taken any other investigational product in last 4 weeks.
4. Patients having untreated symptomatic dental infection.
5. Patients with WHO Grade 3 or 4 oral Mucositis.
6. Other serious concurrent illness.
7. Inconclusive histological diagnosis.
8. Patients on anticancer antibiotics.
9. Patients with signs and symptoms of systemic infections.
10. Patient's/guardian's refusal to sign informed consent.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of mucositis grade(Common Terminology Criteria of Adverse Events (CTCAE) and World health Organization (WHO) | Day 0-Days 24
  1. Determine the incidence of grade III and IV mucositis in patients undergoing allogeneic or autologous haematopoietic stem cell transplantation in two groups

SECONDARY OUTCOMES:
Incidence,duration and time period of mucositis Common Terminology Criteria of Adverse Events (CTCAE) and World health Organization (WHO) | Day 0-Days 24
  1. Determine the incidence of all Grade of mucositis in patients undergoing allogenic or autologous haematopoietic stem cell transplantation in two groups (Criteria for assessment is given in Appendix 1).
Incidence,duration and time period of mucositis Common Terminology Criteria of Adverse Events (CTCAE) and World health Organization (WHO) | Day0- days 24
  Duration of and time period for healing of chemotherapy induced oral mucositis.
Incidence,duration and time period of mucositis Common Terminology Criteria of Adverse Events (CTCAE) and World health Organization (WHO) | day 0- days 24
  Determine incidence and severity of dysphagia and requirement of IV antibiotics in two groups

OTHER OUTCOMES:
Safety assessment | D0-D24
  1 Vital Signs (blood pressure, pulse rate and respiratory rate) 2 Laboratory Examinations 5 Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Atul Sharma, MD,DM, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Institute Rotary Cancer Hospital,All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Sharma A, Rath GK, Chaudhary SP, Thakar A, Mohanti BK, Bahadur S. Lactobacillus brevis CD2 lozenges reduce radiation- and chemotherapy-induced mucositis in patients with head and neck cancer: a randomized double-blind placebo-controlled study. Eur J Cancer. 2012 Apr;48(6):875-81. doi: 10.1016/j.ejca.2011.06.010. Epub 2011 Jul 6. PMID 21741230